CLINICAL TRIAL: NCT05244421
Title: SAY San Diego Dad Corps FIRE Healthy Marriage and Responsible Fatherhood Program Evaluation
Brief Title: SAY San Diego Dad Corps FIRE Program Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Evaluation & Research (Other)
Collaborators: Social Advocates for Youth (SAY) San Diego Dads Corps (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #2021/03/40
Record Dates: First submitted 2022-02-08; First posted 2022-02-17 (Actual); Results first posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Fathers

STUDY DESIGN:
Intervention Model Description: Primary services: Participants receive 16 hours of 24/7 Dads curricula, 4 hours of Healthy Relationships workshops, and 4 hours of Economic Stability workshops over the course of 8 weeks. Participants also receive ongoing job readiness support and post-employment support.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Primary Services (Experimental): Primary services: Participants receive 16 hours of 24/7 Dads curricula, 4 hours of Healthy Relationships workshops, and 4 hours of Economic Stability workshops over the course of 8 weeks. Participants also receive ongoing job readiness support and post-employment support.
  Interventions: Other: Primary Services

INTERVENTIONS:
Other: Primary Services — Primary services: Participants receive 16 hours of 24/7 Dads curricula, 4 hours of Healthy Relationships workshops, and 4 hours of Economic Stability workshops over the course of 8 weeks. Participants also receive ongoing job readiness support and post-employment support.

SUMMARY:
The purpose of the SAY San Diego Dad Corps FIRE program evaluation is to determine whether primary (i.e., behaviors) and secondary (i.e., attitudes) outcomes around parenting, co-parenting, employment, job readiness, and financial stability improve for participants after completing the SAY SDDC FIRE program.

DETAILED DESCRIPTION:
After being informed about the study and giving consent, participants will enroll in an eight-week program that collects data at enrollment, at the end of the program, and 12 months following the program. Research questions in this study are framed by a descriptive evaluation design to assess whether outcomes improve for low-income fathers who participate in the SAY SDDC FIRE program. Primary and secondary outcomes are assessed before and after participants complete core curricula - 24/7 Dads, Healthy Relationships, and Economic Stability workshops (pre to post). Primary outcome measures will indicate whether behaviors improved for healthy family relationships (parent, co-parent, and partner) and economic stability (financial, employment). Secondary outcome measures will indicate whether improvements were made in the attitudes and expectations that facilitate and reflect behavior for healthy partner relationships and financial stability.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age 18 and older)
* Father/father figure
* Has a child under the age of 24
* Reside in the San Diego, CA area

Exclusion Criteria:

* Minor (under the age of 18)
* Not a father/father figure
* Fathers with children over the age of 24
* Reside outside of San Diego, CA area

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Father or father-figure
Enrollment: 444 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2025-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matt D Shepherd, PhD, Principal Investigator — Midwest Evaluation & Research
Locations (1):
- Social Advocates for Youth (SAY San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
All participant data will be confidential and aggregated. No individual participant data will be released unless requested by the courts. This study looks at data as a whole.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Primary Services
Started | 444
Completed | 444
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Primary Services
Number analyzed (Participants) | 444
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 443
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 37.28 [20 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 404
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 13
  Asian | 22
  Native Hawaiian or Other Pacific Islander | 9
  Black or African American | 58
  White | 155
  More than one race | 173
  Unknown or Not Reported | 14

OUTCOME MEASURES:

1. Primary Outcome: Healthy Parenting Behavior Measurement #1
Description: Will participants report significantly healthier parenting behavior after completing primary educational services and employment support services?
  Items measured include:
  Parenting behavior and interaction with children measured with:
  9 items- frequency of engagement in key behaviors (categories, 5-point scale)
  Measured on the Healthy Parenting Behavior Scale #1 as:
  1=Never 2=1 to 2 days per month 3=3 or 4 days per month 4=2 or 3 days per week 5=Every day or almost every day Higher ratings indicate higher frequency of engagement in parenting behavior and interaction with children, so the higher the rating, the better the score.
  The 9 items are measured as a construct. All items are added together and divided by 8 to create the construct score. The higher the score, the better the outcome.
  maximum score of 5.0, minimum score of 1.0
Time Frame: Change from baseline in behavior in parenting behavior (interaction with children at 12 months from enrollment)
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Primary Services
Number analyzed (Participants) | 97
score on scale
  mean at baseline | 3.93 (.900)
  mean at follow-up | 4.26 (.761)

2. Primary Outcome: Healthy Co-parenting Behavior Measurement #1
Description: Will participants report significantly healthier co-parenting behavior after completing primary and employment support services?
  Items measured include:
  Co-parenting behavior measured with:
  11 items: frequency of agreement with key co-parenting behaviors (interval, 5-point scale)
  Measured on the Healthy Co-Parenting Behavior Scale #1 as:
  1. Strongly Disagree
  2. Disagree
  3. Neutral
  4. Agree
  5. Strongly Agree
  The 11 items are measured as a construct. All items are added together and divided by 11 to create the construct score. The higher the score, the better the outcome.
  maximum score of 5.0, minimum score of 1.0
Time Frame: Change from baseline in co-parenting behavior at 12 months from enrollment
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Primary Services
Number analyzed (Participants) | 156
score on scale
  mean at baseline | 3.23 (1.166)
  mean at follow-up | 3.28 (1.171)

3. Primary Outcome: Healthy Financial Behavior Measurement #1
Description: Will participants report significantly healthier financial behavior after completing primary educational employment support services?
  Items measured include:
  Father financial behavior measured with:
  3 items: yes (1) or no (0) questions for have resume, checking account, savings account (dichotomous) Yes (1) responses indicate financial readiness, so the higher the rating, the better the score.
Time Frame: Change from baseline in father financial behavior at 12 months from enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Services
Number analyzed (Participants) | 234
Participants
  Have saving account-baseline | 61
  Have savings account-follow-up | 105
  Have resume-baseline | 56
  Have resume-follow-up | 99
  Have checking account-baseline | 53
  Have checking account-follow-up | 150

4. Secondary Outcome: Healthy Parenting Attitudes Measurement #1
Description: Will participants report significantly healthier parenting attitudes after completing primary educational employment support services?
  Items measured include:
  Parenting attitudes toward children measured with:
  7 items: frequency of key attitudes (categories, 5-point scale)
  Measured on the Healthy Parenting Attitudes Scale #1 as:
  1. Always
  2. Often
  3. Sometimes
  4. Rarely
  5. Never
  The 7 items are measured as a construct. All items are added together and divided by 7 to create the construct score. The higher the score, the better the outcome.
  maximum score of 5.0, minimum score of 1.0.
Time Frame: Change in parenting attitudes (towards children) from baseline to immediately after program completion (8 weeks).
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Primary Services
Number analyzed (Participants) | 158
score on scale
  mean at baseline | 4.45 (.531)
  mean at follow-up | 4.48 (.535)

ADVERSE EVENTS:
Time Frame: 1 year through study completion
Description: The definition of adverse events does not differ from clinicaltrials.gov
Arm/Group | Primary Services
All-Cause Mortality (participants affected / at risk) | 0/444
Serious Adverse Events (participants affected / at risk) | 0/444
Other Adverse Events (participants affected / at risk) | 0/444

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-05-24): https://cdn.clinicaltrials.gov/large-docs/21/NCT05244421/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-24): https://cdn.clinicaltrials.gov/large-docs/21/NCT05244421/SAP_001.pdf